CLINICAL TRIAL: NCT06561958
Title: Prospective, Multi-country, Non-Interventional Study to Investigate REKOVELLE for Ovarian Stimulation: the Effectiveness, Safety, and Patterns Of Use for Asian Women in Real World Practice
Brief Title: Prospective, Multi-centre, Non-Interventional Study to Investigate the Effectiveness of REKOVELLE® for Ovarian Stimulation for Asian Women in Real World Settings
Acronym: PROFOUND
Status: Recruiting | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000430
Record Dates: First submitted 2024-08-06; First posted 2024-08-20 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- REKOVELLE: Participants prescribed REKOVELLE for the first time for controlled ovarian stimulation.
  Interventions: Drug: REKOVELLE

INTERVENTIONS:
Drug: REKOVELLE — Individualised dosing regiment of REKOVELLE in routine clinical practice.

SUMMARY:
Primary objective is to investigate the effectiveness of REKOVELLE® in women undergoing their first REKOVELLE® ovarian stimulation treatment in real world practice in Asian countries.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 20 years or older at enrollment
* Serum AMH level >0.5 ng / mL (with the latest result tested within 12 months)
* Who are first time prescribed REKOVELLE for their ovarian stimulation and IVF or ICSI treatment cycle using fresh or frozen ejaculated sperm from male partner or sperm donor (if applicable)
* Willing and able to provide written informed consent

Exclusion Criteria:

* Have undergone more than 2 COS-IVF / ICSI cycles before the enrollment
* Participating in an interventional clinical trial in which any medication treatment is mandated
* Women with a contraindication for prescription of REKOVELLE treatment
* Oocyte donors
* Undergoing ovarian stimulation for fertility preservation

Min Age: 20 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Approximately 1500 patients prescribed REKOVELLE for the first time for controlled overian stimulation (COS) will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative live birth rate | Up to 12 months
  Cumulative live birth rate defined as delivery of at least 1 live fetus after 20 completed weeks of gestation, combined fresh and frozen embryo transfers within 12 months after the start of the ovarian stimulation in patients of the first REKOVELLE ovarian stimulation cycle.

SECONDARY OUTCOMES:
The Luteinising hormone (LH) surge suppression protocol | Up to 22 days
  Treatment pattern will be measured by analysing the Lutenising hormone (LH) surge suppression protocol.
Daily Dosage | Up to 22 days
  Treatment pattern will be measured by analysing the REKOVELLE and concomitant ovarian stimulation protocols, consisting of daily dosage.
Stimulation Duration | Up to 22 days
  Treatment pattern will be measured by analysing the REKOVELLE and concomitant ovarian stimulation protocols, consisting of stimulation duration.
Total Dosage | Up to 22 days
  Treatment pattern will be measured by analysing the REKOVELLE and concomitant ovarian stimulation protocols, consisting of total dosage.
Trigger Protocol | Up to 22 days
  Treatment pattern will be measured by analysing the trigger protocol.
Luteal phase support protocol | Up to 22 days
  Treatment pattern will be measured by analysing the luteal phase support protocol.
Number of oocytes retrieved | Up to 22 days
  Number of oocytes retrieved at oocyte retrieval
Number of Metaphase II (MII) oocytes | Up to 22 days
  Number of MII oocytes at oocyte retrieval (only applicable for Intracytoplasmic sperm injection (ICSI))
Number of embryos | Day 3 after oocyte retrieval
  Number of embryos on Day 3 after oocyte retrieved
Number of Blastocysts | Day 5 after oocyte retrieval
  Number of Blastocysts on Day 5 after oocyte retrieved
Number of embryos transferred | Up to 28 days
  Embryos transferred in fresh and/or frozen transfer cycles
Number of blastocysts transferred | Up to 28 days
  Blastocysts transferred in fresh and/or frozen transfer cycles
Implantation rate | Up to 28 days
  Number of gestational sacs, embryos or blastocysts transferred
Positive human chorionic gonadotropin (hCG) rate | 11 to 15 days after transfer
  Positive human chorionic gonadotropin (hCG) rate analysed using serum or urine hCG test 11-15 days after transfer
Clinical Pregnancy rate | 4 to 5 weeks after transfer
  Clinical pregnancy rate (at least 1 gestational sac 4-5 weeks after transfer)
Vital Pregnancy | 4 to 5 weeks after transfer
  Vital pregnancy rate (at least 1 intrauterine gestational sac with fetal heartbeat 4-5 weeks after transfer)
Ongoing pregnancy rate | 9 to 11 weeks after transfer
  Ongoing pregnancy rate (at least 1 intrauterine viable fetus 9-11 weeks after transfer)
Time to pregnancy | 4 to 5 weeks after transfer
  Time to pregnancy from start date of ovarian stimulation to confirmation of clinical pregnancy
Live birth rate | More than 20 weeks after transfer
  Live birth is defined as delivery of at least 1 live fetus after 20 completed weeks of gestation within 12 months after the start of the ovarian stimulation in patients of the first REKOVELLE ovarian stimulation cycle.
Multiple pregnancy rate | 4 to 5 weeks after transfer
  More than 1 gestational sac with fetal heart beat 4-5 weeks after transfer
Spontaneous abortion rate | Up to 10-11 weeks after transfer
  Spontaneous abortion is defined as positive hCG test but all intrauterine gestational sacs without fetal heart beat as documented by ultrasound, or there are no viable fetuses observed by ultrasound
Ectopic pregnancy rate | Up to 10-11 weeks after transfer
  Ectopic pregnancy is defined as extrauterine gestational sac with or without fetal heart beat as documented by ultrasound or surgery.
Estradiol Hormone levels | Up to 20 days
  Estradiol hormone levels before stimulation and at the end of stimulation day
Progesterone Hormone levels | Up to 20 days
  Progesterone hormone levels before stimulation and at the end of stimulation day
Cycle cancellation rate and the reason for cycle cancellation | Up to 28 days
  Date when the investigator decides to cancel cycle before oocyte pick up (due to poor ovarian response, excessive ovarian response, any illness which prevents oocyte collection procedure, subject not taking hCG injection at the correct time, subject choice, other) or after oocyte pick-up (due to no oocytes collected, no oocytes fertilized, abnormal fertilization, abnormal embryo development, no embryo development, ovarian hyperstimulation syndrome (OHSS), subject choice, any other specified reason)
Transfer cancellation rate and the reason for transfer cancellation | Up to 28 days
  Transfer cancellation rate and the reason for transfer cancellation (no embryo available for transfer, risk of OHSS, endometrium not receptive, high progesterone level, adverse event, any other specified reason for transfer cancellation).
Frequency and severity of adverse drug reactions (ADRs) and serious adverse events (SAEs) | During 1st cycle with REKOVELLE (each cycle range is 5-20 days, average 9 days), Up to 10-11 weeks after transfer
  Frequency and severity of ADRs and SAEs as defined by the investigator
Preventive interventions for ovarian hyperstimulation syndrome (OHSS) | During 1st cycle with REKOVELLE (each cycle range is 5-20 days, average 9 days), Up to 10-11 weeks after transfer.
  Preventive interventions decided by the investigator (Triggering of final follicular maturation with GnRH agonist and fresh embryo/blastocyst transfer or cryopreservation, Cancellation of fresh embryo/blastocyst transfer)
Number of subjects with mild / moderate / severe ovarian hyperstimulation syndrome (OHSS) | During 1st cycle with REKOVELLE (each cycle range is 5-20 days, average 9 days), Up to 10-11 weeks after transfer
  Number of subjects with mild / moderate / severe OHSS, defined by the investigator

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (27):
- Japan (12):
  - Ferring Investigational Site, Chiba, Chiba
  - Ferring Investigational Site, Fukuoka, Fukuoka
  - Ferring Investigational Site, Kitakyushu, Fukuoka
  - Ferring Investigational Site, Takasaki, Gunma
  - Ferring Investigational Site, Hiroshima, Hiroshima
  - Ferring Investigational Site, Bunkyō City, Japan
  - Ferring Investigational Site, Tokyo, Tokyo
  - Ferring Investigational Site, Hiroshima
  - Ferring Investigational Site, Hokkaido
  - Ferring Investigational Site, Hyōgo
  - Ferring Investigational Site, Osaka
  - Ferring Investigational Site, Saitama
- South Korea (5):
  - Ferring Investigational Site, Busan, Busan
  - Ferring Investigational Site, Daegu, Daegu
  - Ferring Investigational Site, Seongnam-si, Seongnam
  - Ferring Investigational Site, Busan
  - Maria Fertility Hospital, Seoul
- Taiwan (4):
  - Ferring Investigational Site, Tainan, Tainan
  - Ferring Investigational Site, Taoyuan District, Taoyuan
  - Ferring Investigational Site, Taichung
  - Ferring Investigational Site, Taipei
- Thailand (3):
  - Naresuan University Hospital, Phitsanulok, Muang
  - Ramathibodi Hospital, Bangkok, Ratchathewi
  - Ferring Investigational Site, Bangkok
- Vietnam (3):
  - Ferring Investigational Site, Hanoi, Hanoi
  - Ferring Investigational Site, Ho Chi Minh City, Ho Chi Minh City
  - Ferring Investigational Site, Huế, Huế

IPD SHARING:
Plan to Share IPD: No